CLINICAL TRIAL: NCT05551715
Title: Virtual Eye Model System for Personalised Refractive Surgery Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vissum, Instituto Oftalmológico de Alicante (Other)
Collaborators: COSTRUZIONI STRUMENTI OFTALMICI C.S.O. SRL (Unknown); Unidade Local de Saúde de Coimbra, EPE (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jorge Alio, Principal investigator, Vissum, Instituto Oftalmológico de Alicante
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VEMoS
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Individualized Refractive Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Untreated eyes (Other): Participants in the untreated arm will undergo an ophthalmic examination only once.
  Interventions: Device: Software development for individualized refractive surgery
- Refractive surgery (Other): Participants on this arm will undergo two ophthalmic examinations, one before and one after surgery. For refractive surgery participants, refractive surgery will be performed as part of the habitual clinical practice. All other additional tests performed as part of the clinical trial are all non-invasive.
  Interventions: Device: Software development for individualized refractive surgery
- Cataract surgery (Other): Participants on this arm will undergo two ophthalmic examinations, one before and one after surgery. For cataract surgery participants, cataract surgery will be performed as part of the habitual clinical practice. All other additional tests performed as part of the clinical trial are all non-invasive.
  Interventions: Device: Software development for individualized refractive surgery

INTERVENTIONS:
Device: Software development for individualized refractive surgery — Software development for individualized refractive surgery

SUMMARY:
Justification: Although great strides have been made in the past to develop VEMoS software, it has not yet been validated with actual clinical data from patients who have undergone cataract or refractive surgery.

There are some fundamental questions that must be addressed to validate and update the software, such as the objective visual quality metrics that best predict the patient's post-surgical subjective vision from the predictions of the optical properties of the eye.

The VEMoS software must be adjusted for different types of inputs and eye parameters:

Corneal tomography of MS39-AXL MS39-AXL corneal tomography + biometric data from the IOL Master MS39-AXL corneal tomography + IOL Master biometric data + total aberrometry Combinations of any of the above with the optical properties of a specific IOL, etc.

Objective The main objective is to standardize the selection of parameters to personalize refractive surgery, based on the biometric data of each patient.

The objectives necessary to achieve such an ambitious goal are:

1. Redesign VEMoS software
2. Determine which biometric data, diagnostic tools, and objective and subjective metrics of visual quality are best for the selection of optimal refractive parameters for surgery
3. Optimize the combined use of biometric data, VEMoS software, and visual quality metrics Study design The proposed multicenter clinical trial is observational and prospective. There will be three arms within the clinical trial, a no-treatment arm, a refractive surgery arm, and a cataract surgery arm. Participants in the untreated arm will undergo an ophthalmic exam only once. Participants in the other two arms will undergo two ophthalmic exams, one before and one after surgery. For all participants, cataract or refractive surgery will be performed as part of routine clinical practice. Other additional tests performed are all non-invasive.

Study population Untreated eye arm patients 18 to 40 years of age. Refractive surgery arm patients who are planned and have consented to a corneal refractive procedure to gain spectacle independence.

Cataract surgery arm patients older than 50 years who are planned and have consented to cataract surgery.

Sample size The sample sizes for each arm of the clinical trial are as follows.

Untreated eye arm:

The goal is to recruit 600 eyes from 300 patients, 100 patients in each of these groups:

Myopia (from -10 D to -0.75 D) Emmetropia (from -0.5 D to + 0.5 D) Hyperopia (from 0.75 D to 5 D)

Refractive surgery arm:

For LASIK, the goal is to recruit 800 eyes from 400 patients, 100 patients in each of these groups:

High myopia (from -10 D to -6 D) Medium myopia (from -6 D to -3 D) Low myopia (from -3 D to -1 D) Hyperopia (from +1 D to +4 D)

For SMILE, the goal is to recruit 400 eyes from 200 patients, 100 patients in each of these groups:

High myopia (from -10 D to -6 D) Average myopia (from -6 D to -3 D)

For the cataract surgery arm:

The goal is to recruit 400 eyes from 200 patients, 100 patients in each of these groups Zeiss monofocal IOLs multifocal IOL

A total of 500 patients are expected between the Vissum, IMO and IOA clinics in Miranza.

A total of 250 patients are expected between hospital and university of Coimbra epe (Portugal).

A total of 350 patients are expected at Aarhus universitetshospital (Denmark).

ELIGIBILITY:
Inclusion Criteria:

For the untreated eyes arm, the inclusion criterion is:

• patients from 18 to 40 years of age and with less than 2 D of astigmatism.

For the refractive surgery arm, the inclusion criteria are:

* for LASIK: sphere between -10 D and +4 D and with less than 3 D of astigmatism.
* for SMILE: sphere between -10 D and -3 D, with less than 3 D of astigmatism.

For the cataract surgery arm, the inclusion criterion is:

• patients older than 50 years old without any active ocular pathologies affecting visual capabilities except cataract and with less than 1 D of astigmatism.

Exclusion Criteria:

For the untreated eyes and the refractive surgery arms, the exclusion criteria are:

* ocular pathology affecting visual capabilities,
* reduced transparency of ocular media,
* systemic disease affecting visual capabilities.

For the cataract surgery arms, the exclusion criterion is:

* Systemic disease affecting visual capabilities.
* Ocular pathology affecting visual capabilities other than cataract
* Included patients will be excluded if surgical complications occurs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 547 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Variables to run the VEMoS software and obtain estimates and simulations Corneal Topography | 3 months
  To evaluate the keratomery in diopters
Variables to run the VEMoS software and obtain estimates and simulations Pupil size | 3 months
  To evaluate pupil size at different illumination in milimeters
Variables to run the VEMoS software and obtain estimates and simulations anterior chamber depth | 3 months
  To obtain the anterior chamber depth in milimeters
Variables to run the VEMoS software and obtain estimates and simulations, crystalline lens thickness | 3 months
  To obtain the crystalline lens thickness in milimeters
Variables to run the VEMoS software and obtain estimates and simulations, axial length | 3 months
  To obtain the axial length in milimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Alicante Vissum Miranza, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No